CLINICAL TRIAL: NCT02210234
Title: Wheat Bioactives and Immune Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Kellogg's Corporate Citizens Fund (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 114-2010
Record Dates: First submitted 2014-08-05; First posted 2014-08-06 (Estimated); Last update posted 2014-08-06 (Estimated); Status verified 2014-08

CONDITIONS: Endocrine, Nutritional, Metabolic and Immunity Disorders
Keywords: wheat bran; healthy immunity; T cells
MeSH Terms: conditions — Immune System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 50 grams of whole wheat bran cereal (Active Comparator): This arm was randomized to eat 50 grams of whole wheat brand cereal during the day for 3 weeks.
  Interventions: Dietary Supplement: 50 grams of whole wheat bran cereal
- 100 grams of whole wheat bran cereal (Active Comparator): This arm was randomized to eat 100 grams of whole wheat brand cereal the day for 3 weeks.
  Interventions: Dietary Supplement: 100 grams of whole wheat bran cereal

INTERVENTIONS:
Dietary Supplement: 50 grams of whole wheat bran cereal — This arm was randomized to eat 50 grams of whole wheat cereal during the day for 3 weeks. At baseline and at week 3 a blood sample was taken to determine if there was any alteration to the proliferation of gamma-delta T-cells.
  Other Names: Kellogg's brand whole wheat bran cereal
  Arms: 50 grams of whole wheat bran cereal
Dietary Supplement: 100 grams of whole wheat bran cereal — This arm was randomized to eat 100 grams of whole wheat cereal during the day for 3 weeks. At baseline and at week 3 a blood sample was taken to determine if there was any alteration to the proliferation of gamma-delta T-cells.
  Other Names: Kellogg's brand whole wheat bran cereal
  Arms: 100 grams of whole wheat bran cereal

SUMMARY:
The purpose of this research was to understand the effects of bioactive compounds found in wheat cereal on human immunity. Subjects came in for a baseline blood draw, consumed whole wheat bran cereal daily for 21 days, and returned for a final blood draw. Immune function assays were performed at both sampling times. It was predicted that eating wheat bran would benefit immune function.

DETAILED DESCRIPTION:
Healthy individuals, between 18 and 50 years of age, were recruited by flyer and word of mouth on the University of Florida campus and in the surrounding area, in May of 2010. Eligible subjects were randomly assigned to one of two experimental groups, to consume either 50 grams or 100 grams of whole wheat bran cereal daily, for three weeks. Blood was drawn from fasting subjects before consumption (baseline) and after three weeks of cereal consumption. Peripheral blood mononuclear cells (PBMC) were isolated and cultured with a broad based mitogen and autologous serum for 10 days. PBMC were stained with fluorochrome-conjugated antibodies on Day 0 and Day 10 of culture, at each blood draw. Data was acquired by flow cytometry and analyzed. Overall compliance was assessed using self-reported data and by counting left-over bags of cereal.

ELIGIBILITY:
Inclusion Criteria:

* generally healthy
* aged 18-65

Exclusion Criteria:

* chronic health problems
* high blood pressure
* BMI greater than 25
* vegan

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2010-05; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
γδ-T cell proliferation | Change in Baseline and 3 weeks
  Flow cytometry is used to compare the percentage of γδ-T cells in the total CD3 cell population in the blood of subjects before and after three weeks of consuming whole wheat bran cereal. An increase in that percentage would be suggestive of improved immunity (priming).

CONTACTS AND LOCATIONS:
Overall Officials: Susan S Percival, PhD, Principal Investigator — University of Florida
Locations (1):
- Department of Food Science & Human Nutrition, University of Florida, Gainesville, Florida, United States